CLINICAL TRIAL: NCT00959959
Title: ARMOR1: Phase 1, Open Label, Dose Escalation Trial of TOK-001 for the Treatment of Chemotherapy Naive Castration Resistant Prostate Cancer
Brief Title: ARMOR1: Study of TOK-001 to Treat Castration Resistant Prostate Cancer
Acronym: ARMOR1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LTN PHARMACEUTICALS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOK-200-05
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: CRPC; HRPC; TOK-001; ARMOR; ARMOR1; ESL; Galeterone
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 650 mg TOK-001 (Experimental)
  Interventions: Drug: TOK-001
- 1300 mg TOK-001 (Experimental)
  Interventions: Drug: TOK-001
- 1950 mg TOK-001 (Experimental)
  Interventions: Drug: TOK-001
- 975 mg TOK-001 (Experimental)
  Interventions: Drug: TOK-001
- 975 mg TOK-001, supplement (Experimental)
  Interventions: Drug: TOK-001
- 1950 mg TOK-001, split dose (Experimental)
  Interventions: Drug: TOK-001
- 2600 mg TOK-001 (Experimental)
  Interventions: Drug: TOK-001
- 2600 mg TOK-001, split dose (Experimental)
  Interventions: Drug: TOK-001

INTERVENTIONS:
Drug: TOK-001 — 2 capsules (325 mg each), once per day
  Other Names: Dose Group 1
  Arms: 650 mg TOK-001
Drug: TOK-001 — 4 capsules (325 mg each), once per day
  Other Names: Dose Group 3
  Arms: 1300 mg TOK-001
Drug: TOK-001 — 6 capsules (325 mg each), once per day
  Other Names: Dose Group 4
  Arms: 1950 mg TOK-001
Drug: TOK-001 — 3 capsules (325 mg each), once per day
  Other Names: Dose Group 2
  Arms: 975 mg TOK-001
Drug: TOK-001 — 3 capsules (325 mg each), once per day with supplement
  Other Names: Dose Group 5
  Arms: 975 mg TOK-001, supplement
Drug: TOK-001 — 6 capsules (325 mg each), split dose (3 capsules with breakfast, 3 capsules with dinner)
  Other Names: Dose Group 6
  Arms: 1950 mg TOK-001, split dose
Drug: TOK-001 — 8 capsules (325 mg each), once per day
  Other Names: Dose Group 7
  Arms: 2600 mg TOK-001
Drug: TOK-001 — 8 capsules (325 mg each), split dose (4 capsules with breakfast, 4 capsules with dinner)
  Other Names: Dose Group 8
  Arms: 2600 mg TOK-001, split dose

SUMMARY:
The purpose of this study is to determine whether TOK-001 is safe and shows biological effect in the treatment of castration resistant prostate cancer (CRPC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Confirmed cancer of the prostate
* Progressing disease in spite of androgen ablation therapy
* Able to swallow multiple capsules

Exclusion Criteria:

* Participation in another clinical trial < 4 weeks prior to enrollment
* Metastatic disease with one or more of the following:

  * Liver involvement
  * Bone pain associated with confirmed evidence of metastases
  * Non-hepatic visceral involvement
* The following medications:

  * Prior treatment with MDV3100, abiraterone, Provenge or TAK700
  * Prior treatment with ketoconazole
  * Prior treatment with chemotherapy
  * Prior radiation therapy completed ≤ 4 weeks prior to enrollment
* The following medical conditions:

  * Active angina pectoris
  * History of Hepatitis B or Hepatitis C
  * Known HIV infection
  * Ongoing hypertension

Note: There are additional inclusion and exclusion criteria. The clinical site center will determine if you are eligible. If you are not eligible for the trial, site staff will detail the reasons to you.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Phase 1: Incidence of adverse events | 3 months
  Safety will be assessed by incidence of AEs and change from baseline in the following additional safety parameters: clinical laboratory assessments, physical examination, vital signs, and 12 lead electrocardiograms (ECGs)

SECONDARY OUTCOMES:
Efficacy Measures | 3 months
  Efficacy will be assessed by evaluation of change in PSA level, changes from baseline in CT/MRI and bone scans, response rate RECIST criteria and additional special laboratories

CONTACTS AND LOCATIONS:
Overall Officials: R. B. Montgomery, MD, Principal Investigator — University of Washington; M. E. Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada & US Oncology Research, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington